CLINICAL TRIAL: NCT01120756
Title: Neural Bases of Cognitive Rehabilitation for Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B7467-I
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Brain Injury
Keywords: executive dysfunction; brain injury; attention; rehabilitation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Goal-oriented attentional self-regulation training (Experimental): Goal-oriented attentional self-regulation training (GOALS).
  Interventions: Behavioral: Goal-oriented attentional self-regulation
- Brain Health Education (Active Comparator): Brain Health Education (EDU)
  Interventions: Behavioral: Brain Health Education

INTERVENTIONS:
Behavioral: Goal-oriented attentional self-regulation — This will involve 5-7 weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training (1 hour at the beginning, halfway through and at the end of training), and approximately 20 hours of home practice). In brief, the GBSM training protocol is designed to maximize the potential for improving attention regulation skills and the goal-directed functions they support, applying mindfulness-based attention regulation training to practice in redirecting attention to goal-relevant processes especially in the context of distractions is emphasized throughout training. Participants are asked to identify realistic functional goals as feasible individual and group projects, and are then trained in goal management strategies on the functional task(s) of their choice.
  Arms: Goal-oriented attentional self-regulation training
Behavioral: Brain Health Education — Brain Health Education (EDU) will involve 5-7 weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training (1 hour at the beginning, halfway through and at the end of training), and approximately 20 hours of homework). The EDU intervention involves education in health and brain injury in a classroom format, with study materials for homework.
  Arms: Brain Health Education

SUMMARY:
Some of the most common and disabling consequences of brain injury are deficits in cognition, such as difficulty with sustained attention, memory, organization, and goal management. The long-term goal of this research program is to develop and test novel neuroscience-based cognitive interventions for improving attentional regulation and related "executive function" brain processes involved in goal-directed behavior.

DETAILED DESCRIPTION:
Brain injury often results in a disruption of attention regulation processes, which reduces the efficiency and effectiveness of cognitive functions including learning, memory, problem-solving and goal management, leading to significant functional disability. More intervention options are needed.

We set out to test different possible interventions. Individuals with traumatic brain injury (TBI) and chronic executive control dysfunction participate in interventions, with pre- and post-intervention measurements of cognitive functioning. Training in Goal-oriented attentional self-regulation (GOALS) was administered in comparison to Brain Health Education (EDU).

GOALS is designed to train attention regulation skills along with meta-cognitive strategies for goal management, with a emphasis on application to participant-selected projects. This is a group-based intervention.

Brain Health Education is designed to increase knowledge and understanding of key factors that affect brain functioning. This is a group-based intervention matched to the GOALS intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients with a history of TBI (reported plausible mechanism of head injury, loss of consciousness with some period of post-traumatic alteration in cognition) who are > 6 months post-injury will be screened for evidence of mild-moderate residual dysfunction in executive control functions based on corroborated reports of real-world difficulties (Mayo-Portland Adaptability Inventory).

Exclusion Criteria:

* Severely apathetic/abulic
* aphasic
* or other reasons for patients being unable or unwilling to participate with the training tasks
* severe cognitive dysfunction
* history of neurodevelopmental abnormalities
* ongoing illicit drug or alcohol abuse (AUDIT>8)
* severe depression as measured by Beck Depression Inventory (>29)
* severe PTSD precluding participation in research activities (such as group training or MRI scanning)
* There will be no restriction in regard to gender, race and socioeconomic status.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Chen, MD MA, Principal Investigator — Martinez Outpatient Clinic, Martinez, CA
Locations (1):
- Martinez Outpatient Clinic and Community Living Center, Martinez, CA, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Novakovic-Agopian T, Kornblith E, Abrams G, Burciaga-Rosales J, Loya F, D'Esposito M, Chen AJW. Training in Goal-Oriented Attention Self-Regulation Improves Executive Functioning in Veterans with Chronic Traumatic Brain Injury. J Neurotrauma. 2018 Dec 1;35(23):2784-2795. doi: 10.1089/neu.2017.5529. Epub 2018 Jul 23. PMID 29717652

RESULTS

PARTICIPANT FLOW:
Groups:
- Goal-oriented Attentional Self-regulation Training: Goal-oriented attentional self-regulation training (GOALS).
  This will involve 5-7 weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training (1 hour at the beginning, halfway through and at the end of training), and approximately 20 hours of home practice). In brief, the GBSM training protocol is designed to maximize the potential for improving attention regulation skills and the goal-directed functions they support, applying mindfulness-based attention regulation training to practice in redirecting attention to goal-relevant processes especially in the context of distractions is emphasized throughout training. Participants are asked to identify realistic functional goals as feasible individual and group projects, and are then trained in goal management strategies on the functional task(s) of their choice.
Period: Overall Study
Arm/Group | Goal-oriented Attentional Self-regulation Training | Brain Health Education
Started | 21 | 14
Completed | 20 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Goal-oriented Attentional Self-regulation Training | Brain Health Education | Total
Number analyzed (Participants) | 21 | 14 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (11) | 43 (11) | 43 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on a Composite Measure (Z-score) of Attention, Working Memory, and Executive Functions
Description: We computed a composite measure based upon the average of individuals' scores on commonly used neuropsychological tests of attention, working memory, and executive functions. To compute this composite score, we first scored individual performances on each neuropsychological measure utilizing published norms, adjusted for, when available, age, gender, ethnicity, and education levels. We then converted all resultant scores (e.g., T-scores, Standard Scores) to a common metric, z-scores. (Z-scores are a standardized unit of measurement, scaled in terms of standard deviation (SD) units. Thus, a z-score of 0 represents the mean; a z-score of 1 represents+1 SD above the mean; and a z-score of -1 represents -1 SD below the mean.) Finally, for each participant, z-scores derived from each separate neuropsychological test were averaged together to yield a final composite score. The composite score was the unit of analysis.
Time Frame: Baseline, Within 2-3 weeks Post-intervention
Population: We lost a total of n=2 participants to attrition from baseline to follow-up. This included n=1 from the Goal-Oriented Attentional Self-regulation training and n=1 from the Brain Health Education.
Measure: Mean (Standard Deviation); unit: Change to Z (composite) score
Arm/Group | Goal-oriented Attentional Self-regulation Training | Brain Health Education
Number analyzed (Participants) | 20 | 13
Change to Z (composite) score | 0.26 (.27) | .01 (.25)

2. Secondary Outcome: Functional Evaluations: Change From Baseline on the Goal Processing Scale
Description: Observed measures of functional performance on complex tasks were assessed for the GOALS and Brain Health Education study. The overall composite score comprises scores for planning, initiation, self-monitoring, maintenance of attention, sequencing and switching, divergent thinking, execution, learning and memory. Scores range from 1-10. Changes were calculated from pre-to post-training, and higher scores indicate improvement in functioning.
Time Frame: Baseline, 2-3 Weeks Post-intervention
Population: This measurement was used for the comparison of Goal-oriented attentional self-regulation training and Brain Health Education interventions. Also, we lost a total of n=2 participants to attrition from baseline to follow-up. This included n=1 from the Goal-Oriented Attentional Self-regulation training and n=1 from the Brain Health Education.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Goal-oriented Attentional Self-regulation Training | Brain Health Education
Number analyzed (Participants) | 20 | 13
units on a scale | 1.05 (1.15) | .01 (0.25)

ADVERSE EVENTS:
Time Frame: 6-12 weeks
Arm/Group | Goal-oriented Attentional Self-regulation Training | Brain Health Education
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/14
Other Adverse Events (participants affected / at risk) | 0/21 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT01120756/Prot_SAP_000.pdf